CLINICAL TRIAL: NCT01361841
Title: Effects of Latanoprost, Bimatoprost and Travoprost in Patients With Latanoprost-resistant Glaucoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Responsible Party: Centre Hostitalier Universitaire de Sherbrooke, CHUS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUS-09-184
Record Dates: First submitted 2011-05-25; First posted 2011-05-27 (Estimated); Last update posted 2011-05-27 (Estimated); Status verified 2010-12

CONDITIONS: Ocular Hypertension; Primary Glaucoma
Keywords: Latanoprost; bimatoprost; travoprost; non responders
MeSH Terms: conditions — Ocular Hypertension | interventions — Latanoprost; Bimatoprost; Travoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ophtalmic solution, (Other): Travoprost, latanoprost and bimatoprost, ophthalmic solution are topical medications used for controlling the progression of glaucoma or ocular hypertension, by reducing intraocular pressure. they are synthetic prostaglandin F 2α analogue (and prodrug for bimatoprost) that works by increasing the outflow of aqueous fluid from the eyes.
  Interventions: Drug: Latanoprost, bimatoprost, travoprost; Drug: travoprost, latanoprost and bimatoprost

INTERVENTIONS:
Drug: Latanoprost, bimatoprost, travoprost — topic drops, once a day at bedtime, for years
  Other Names: Xalatan; Lumigan; Travatan
Drug: travoprost, latanoprost and bimatoprost — one drop once a day for life
  Other Names: Travatan; Xalatan; Lumigan

SUMMARY:
Intraocular pressure (IOP) is considered to be the main risk factor for progression of glaucoma and therefore the main target of therapy. Pharmacologic treatment of glaucoma has changed considerably during the last decades due to the introduction of prostaglandin analogues. Three of these are commonly used in North America: latanoprost (Latanoprost T, Pfizer), Travoprost (Travatan TM, Alcon) and bimatoprost (Lumigan TM, Allergan).

There have been several studies to evaluate their effectiveness. The three seem to be equivalent, according to the only study that has compared the molecules. Latanoprost is employed initially, due to its paucity of side effects when compared to the other two analogues. However, if it is not effective, several studies ahve shown that a result is possible using either travoprost or bimatoprost. No study has been conducted to date systematically comparing the three molecules in cases of resistance to latanoprost. In actuality, the investigators patients will receive treatment identical to current practice with the exception of the group continuing with latanoprost. Several studies confirm the benefit of changing prostaglandin analogues if the first has not signficantly decreased the IOP (Palmberg et al. 2004). Each prostaglandin has unique properties which may cause the mechanism of action to vary slightly among patients. (cf. Pharmacological Aspects)

The goal of the study is thus to evaluate the efficaciousness of latanoprost, bimatoprost and travoprost in their IOP-lowering capacity in patients who do not initially respond to latanoprost.

DETAILED DESCRIPTION:
Research question:

What is the effectiveness of latanoprost, bimatoprost and travoprost in patients whose intraocular pressure does not decrease by at least 20% while undergoing treatment with latanoprost ?

Secondary questions:

1- What is the percentage of glaucoma patients who are resistant to latanoprost ? 2- Which prostaglandin is the most effective in decreasing intraocular pressure in cases of resistance to latanoprost ?

Research Project Goals :

Evaluation of the effectiveness of latanoprost, bimatoprost and travoprost in patients in whom latanoprost does not decrease the intraocular pressure by at least 20%. The effectiveness of the three prostaglandins will be determined by the IOP : the treatment should at least effect a 20% decrease from baseline (IOP measured at time of recruitment), with the ultimate aim of attaining the target IOP, which varies depending on the patient. Target IOP is based on the severity of optic nerve damage as well as baseline IOP.

Determine the percentage of patients resistant to prostaglandins. Patients who have not responded (as measured by IOP decrease) to more than 2 prostaglandins will be considered resistant to this category of hypotensive medications.

Study design:

Randomised, open label.

Study duration:

Approximately two years.

POPULATION:

The target population consists of open angle glaucoma patients, or patients with ocular hypertension with an IOP greater than 21 mmHg and who have never undergone treatment for glaucoma. Patients must be 18 years or older, capable of giving informed consent in written form.

Sampling

* Candidates will be selected from the patient population of the ophthalmology clinic of the CHUS hotel-Dieu or from the private practice of Dr. Blondeau
* The patients will all be treated with latanoprost for approximately 6 weeks, after which only those who have not experienced at least a 20% decrease in their initial IOP and who are eligible will be invited to participate in the study.

Sample size - The sample size estimate is based on the need to obtain a significant decrease from baseline IOP at 6 weeks, 2 months and 6 months. Estimating a maximum IOP variation of 2 mmHg with a standard deviation of +/- 2 mmHg, the necessary sample size to power the study (90% with a p < 0.05 using a paired-samples Student T test) is about 47 patients per group.

Methods of randomization and sample make-up:

The study will be a randomized and comparative trial taking place over a period of 12 months. Patients will be distributed by random lots of 6 (ACBCAB, etc) into 3 different groups after a documented non-response (IOP decrease of less than 20%) to latanoprost. Group 1 will remain on Latanoprost 0.005%, Group 2 will switch to travoprost 0.004% and Group 3 will switch to bimatoprost 0.03%. The dose of each medication will be 1 drop daily HS, which is the usual dose in ophthalmological practice and in the scientific literature.

Intraocular pressure will be measured in the same manner for all patients by applanation tonometry.

Thus, for each study participant:

Time of IOP measurement IOP value (mmHg) At time of recruitment 6 weeks after 2 months after 6 months after

* Therefore, 3 groups of patients will have the same measurements taken.

Stages of the study:

1. Patient recruitment:

   - Diagnosis of glaucoma de novo in the outpatient clinic or Dr. Blondeau's office.

   - Patients will be informed about the possibility of resistance to a treatment of 6 weeks with latanoprost, as well as to its possible benefit. The patient will receive a consent form, consisting of an explanation of the study including potential side effects of the medications. Patients will be able to take the time to thoroughly read the document and to decide whether they wish to participate in the study.
2. Consent:

   - Informed consent will be obtained by ophthalmologist Dr. Pierre Blondeau or the resident in ophthalmology, Zineb Ghali, PGY IV, who will offer clarification and explanation to the potential participants if necessary.
3. Trial Design:

1. Patients with a diagnosis of primary open-angle glaucoma (POAG) or ocular hypertension (OH) but who have never received treatment will be recruited.

2. Recruited patients will be treated for 6 weeks with latanoprost. This corresponds to the time necessary for the molecule to block the all prostaglandin receptors, thus allowing for maximum IOP-lowering potential. This period of time was determined by the pharmaceutical company that created the molecule and is used by all studies involving the molecule.

3. Patients who have not experienced a decrease of at least 20% of their baseline IOP and who consent to participate will be distributed into 3 different groups (recruitment step). Group 1 patients will continue to receive latanoprost 0.005%, 1 drop daily HS. The two other groups will receive either bimatoprost 0.03% or travoprost 0.004%, 1 drop daily HS. Patients will continue to be treated for 4 weeks. Patients will receive instructions regarding medication administration and compliance. The medication will be administered every 24 hours between 20:00 and 22:00. No other IOP-lowering medication will be permitted.

4. Patients with less than 20% response to initial treatment with latanoprost will be randomised into 3 groups corresponding to one of the prostaglandin analogues. IOP will be remeasured after 6 weeks in order to evaluate response to the medication. We consider that a documented response to treatment consists of a significant decrease in IOP as measured by the t-test. If the IOP has not decreased by at least 20% after 1 month of treatment with the various prostaglandins, the patient will be excluded from the study, treated with another class of hypotensive agent, and receive standard follow-up.

Security measures:

The researchers will monitor for possible side effects and other potential problems. To this effect, an auxiliary researcher (not yet recruited) as well as a resident in ophthalmology (Zineb Ghali) will be available 24 hours a day to address medication side effects or unexpected symptoms. If immediate follow-up is required and the patient makes contact during business hours, the research team will immediately see the patient. If the patient contacts the auxiliary researcher or the resident outside of business hours, he or she will be immediately referred to one of the ophthalmology residents on call at the hotel Dieu hospital Emergency Department. If necessary, one of the two physician researchers will be available to meet with the patient in question.

This ensures that any adverse reaction will be rapidly treated by the research team. If a physician observes undesirable side effects that are attributable to the medication, he or she has the duty to discontinue treatment as well as the subject's participation in the study. In this case, the physician will ensure continuity of care via another form of treatment in order to ensure the patient's recovery.

Principal dependent variable:

Intraocular pressure shall be measured with a Goldmann tonometer.

A drop of fluorescein sodium and benoxinate hydrochloride, USP (0.25%/0.4%) will be instilled in the patient's eyes, after which baseline IOP will be measured by Goldmann tonometry. The inter-measurement variability is +/- 2mmHg.

Secondary variables:

* Patient age: quantitative
* Patient sex: qualitative
* Patient race: qualitative
* Side effects

  4- Results analysis

Homogeneity of groups in terms of social demographics will be verified via one-way analysis of variance (ANOVA) with Turkey's correction for continuous variables and a chi-square or Fisher's exact test for categorical variables. Values discovered to be significant will be expressed in the following format: obtained value as well as confidence interval, in order to highlight the impact of the particular treatment

Two-way crossed ANOVA will be used to compare data collected during follow-up with different ophthalmological exams, notably the IOP. We will calculate the impact for each period of follow-up.

The incidence of individual side effects will be summarized and compared with a chi-square test. Emphasis will be placed on the degree of severity of symptoms caused by the medications used. The examined side effects will be those that occur most frequently and are of ocular nature.

There is no interim analysis included in this research project. All statistical tests will consider a p-value of less than 0.05 to be statistically significant, i.e. all results will be considered statistically significant at the 5% level.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with ocular hypertension or primary open-angle glaucoma who have never received treatment.
* Age 18 or older and able to give informed consent

Exclusion Criteria:

* Patients with intraocular inflammation of any etiology
* Patients with advanced glaucoma, defined by severe optic nerve damage and/or visual field deficit.
* Patients having had intraocular surgery in the last 4 weeks
* Patients undergoing treatment with ophthalmic solution of any kind
* Patients unable to give informed consent to participate in the research project,including those suffering from psychiatric illness resulting in impaired judgement
* Monophthalmia or anophthalmia
* Pregnant or nursing patients
* Patients status post ocular surgery, with the exception of cataract extraction surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2009-01; Primary Completion 2012-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
intraocular pressure | 2 years
  A drop of fluorescein sodium and benoxinate hydrochloride, USP (0.25%/0.4%) will be instilled in the patient's eyes, after which baseline IOP will be measured by Goldmann tonometry. The inter-measurement variability is +/- 2mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Blondeau, MD, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Locations (1):
- Centre hospitalier de Sherbrooke, Sherbrooke, Quebec, Canada